CLINICAL TRIAL: NCT02594514
Title: Laparoscopic Sleeve Gastrectomy in Severely Obese Adolescents: Effective for Resolution of Cardiovascular Comorbidities
Brief Title: Laparoscopic Sleeve Gastrectomy in Severely Obese Adolescents: Effects on Metabolism
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ruth Rocha Franco, MD, University of Sao Paulo General Hospital
Other Study IDs: USaoPauloLSG
Record Dates: First submitted 2015-10-09; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Obesity; Surgery
Keywords: cardiovascular risk; metabolic profile
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
Severe obesity (SO), defined as BMI≥95th percentile, has increased worldwide among adolescents. American studies estimated that 1.3-2.8% of 12-19-year-old individuals have a BMI >40 kg/m2 or a BMI >35 kg/m2 with at least one serious co-morbidity. The immediate and long-term risks associated with SO in adolescents include cardiovascular and metabolic diseases, obstructive sleep apnoea and nonalcoholic fatty liver disease. However, the results of sleeve gastrectomy in adolescents are still uncertain.

Objective and hypotheses: Investigators aimed to assess the long-term safety, efficacy, and cardiovascular risk changes of laparoscopic sleeve gastrectomy in adolescents with SO.

Method: Longitudinal retrospective study of 22 adolescents with SO who underwent laparoscopic sleeve gastrectomy. Clinical and metabolic variables immediately before surgery and after 6, 12, 18 and 24 months were assessed.

ELIGIBILITY:
Inclusion Criteria:

* ages of 14 and 19
* submitted to LSG between 2007 and 2014.
* attended the child obesity clinic of the pediatric endocrinology department of the Instituto da Criança da Universidade de São Paulo (Children's Institute of University of São Paulo).
* received clinical and pharmacological treatment for at least 6 months before surgery and were followed by a multidisciplinary team including a pediatric endocrinologist, a nutritionist, a psychologist and a physical educator.
* BMI > 40 kg/m2 or BMI > 35 kg/m2 with comorbidities and failed to achieve significant weight loss (10% of initial weight at 6 months) through clinical treatment.
* Both the patients and their guardians were informed about the risks and benefits of surgery and provided informed consent.

Exclusion Criteria:

* it was a retrospective study

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Severe obese adolescents who underwent laparoscopic sleeve gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percent of loss of excess weight following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  weight
percent of reduction in body mass index following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  weight and stature

SECONDARY OUTCOMES:
Changes in insulin resistance following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  laboratory assessment- fasting insulinemia
Changes in total cholesterol and and fractions following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  laboratory assessment-
Changes in glucose and and fractions following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  oral glucose tolerance test
Changes in transaminases following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  laboratory assessment-
Changes in uric acid following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  laboratory assessment-
Changes in triglycerides following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  laboratory assessment-
Changes in abdominal ultrasonography ( steatosis )following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  abdominal ultrasonography
Changes in echocardiogram ( concentric hypertrophy of left ventricle )following laparoscopic sleeve gastrectomy in severely obese adolescents | up to 24 months
  echocardiogram

CONTACTS AND LOCATIONS:
Locations (1):
- HCFUMSP, São Paulo, São Paulo, Brazil